CLINICAL TRIAL: NCT00502099
Title: Phase 4 Comparative Study of Pegasys vs Peg-Intron for Treatment of Chronic Hepatitis C Genotype 4
Brief Title: Comparison of Pegasys Versus Peg-Intron for Treatment of Chronic Hepatitis C Genotype 4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amr Hafez (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Amr Hafez, Doctor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG161190-06
Record Dates: First submitted 2007-07-15; First posted 2007-07-17 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C
Keywords: Chronic hepatitis C; pegylated interferon alfa-2a; ribavirin, rapid virologic response; early virologic response; sustained virologic response
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pegylated interferon alpha 2a plus ribavirin
  Interventions: Drug: Pegylated interferon alpha 2a; Drug: Ribavirin
- 2 (Active Comparator): Pegylated interferon alpha 2b plus ribavirin
  Interventions: Drug: Pegylated interferon alpha 2 b plus ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alpha 2a — Injections: 180 ug once per week
  Other Names: Pegaesys
  Arms: 1
Drug: Ribavirin — Tablets, 1000-1200 daily
  Other Names: Viracure
  Arms: 1
Drug: Pegylated interferon alpha 2 b plus ribavirin — Pegylated interferon alpha 2 b injections
  Other Names: PEG-Interon
  Arms: 2

SUMMARY:
Genotype 4 hepatitis C virus is the cause of approximately 20% of the 170 million cases of chronic hepatitis C in the world. Although rare in western nations, genotype 4 is the most common variant of the hepatitis C virus in Egypt and is also found throughout Africa and the Middle East. Early reports on the treatment of patients with genotype 4 chronic hepatitis C with interferon-alfa (IFN)-alfa monotherapy indicate poor rates of sustained viral response (SVR). With the introduction of ribavirin combination therapy and with pegylation of the IFN alfa molecule, however, response rates have improved dramatically, and current clinical trial data indicate that SVR rates between 43 and 79% are attainable in genotype 4 patients who are receiving pegylated IFN alfa plus ribavirin for 48 weeks. Clinical advances to optimize treatment for each patient have also been made, and tailored treatment options are now being developed that are comparable to the treatment approaches for genotype 1, 2, and 3 patients. A treatment duration of between 36 and 48 weeks appears to be optimal for most patients with chronic hepatitis C genotype 4.The aim of this study is to assess the efficacy and safety of pegylated interferon alpha 2a in patients with chronic hepatitis C genotype 4 in comparison to a historical cohort of patients treated with pegylated interferon alpha 2b

DETAILED DESCRIPTION:
The treatment of chronic hepatitis C with interferon (IFN)-based medicines has advanced steadily since publication of the first clinical trials in the late 1980s.Initial interventions using IFN-alfa monotherapy achieved limited success, but the introduction of IFN-alfa plus ribavirin combination therapy and the pegylation of the IFN alfa molecule, which improved pharmacokinetics and simplified dosing regimens, resulted in a steady improvement in overall treatment outcomes. Sustained virologic responses (SVR, defined as undetectable HCV RNA 24 weeks after completing treatment) have increased from 6% with IFN alfa monotherapy to more than 50% with pegylated interferon alfa (PEG-IFN alfa) plus ribavirin regimensObservations specific to genotype 4 chronic hepatitis C have followed a similar path, with initial investigations of IFN-alfa monotherapy producing limited success .These studies found that IFN-alfa monotherapy, which is usually administered at a dose of 3-5 MIU three times a week for six months, resulted in an SVR in only 5-25% of treated patients.[24-26] The subsequent inclusion of ribavirin in treatment regimens had a dramatic improvement on SVR attainment, with rates of 8 and 42% reported for patients receiving IFN-alfa alone and in combination with ribavirin (1000-1200 mg/day), respectively.

Pegylation of the IFN alfa molecule was the next major advance in the treatment of genotype 4 chronic hepatitis C.Although two early studies failed to demonstrate a significant difference in SVR rates between PEG-IFN alfa-2b plus ribavirin and native IFN alfa-2b plus ribavirin (e.g., 42.9% vs. 32.3%, p = 0.43)[27], subsequent investigations reported SVR rates of 50 to 79% in patients receiving PEG-IFN alfa-2b plus ribavirin (800-1,200 mg/day) for 48 weeks.[ Overall, meta-analysis of clinical trial data shows that SVR rates are significantly higher among genotype 4 patients receiving PEG-IFN alfa plus ribavirin than in those receiving IFN-alfa plus ribavirin (55% vs. 30%, p = 0.0088).[33] This analysis also confirms the importance of adequate ribavirin dosing with higher SVR rates in patients receiving PEG-IFN alfa in combination with high-dose (1000¬-1200 mg/day) and low-dose (800 mg/day) ribavirin (72.0 and 45.8%, respectively; p value not presented). The importance of ribavirin dosing in genotype 4 patients with chronic hepatitis C is also demonstrated in an analysis of the genotype 4 patients included in the registration studies for PEG-IFN alfa-2a.[22, 34] In this analysis, SVR rates were 79% among patients receiving PEG-IFN alfa-2a (180 mcg/week) plus ribavirin (1000-1200 mg/day) for 48 weeks compared with 63% in those receiving the same regimen plus a lower dose of ribavirin (800 mg/day).The optimization of treatment duration is critical in ensuring that SVR rates are maximized without exposing the patient to an unnecessarily long treatment regimen that may have unfavorable implications in terms of cost and tolerability. The question of optimal treatment duration for genotype 4 chronic hepatitis C was addressed in a prospective randomized study in which patients received PEG-IFN alfa-2b (1.5 mcg/kg/week) plus ribavirin (1000-1200 mg/day) for 24, 36, or 48 weeks.Overall, SVR rates were significantly higher in patients receiving treatment for 36 or 48 weeks than in those treated for 24 weeks (66 and 69% vs. 29%; p = 0.001 for each comparison) (Fig. 2). Relapse appeared to be a major factor in determining treatment outcomes: virologic relapse during follow-up was highest among patients treated for 24 weeks (20 of 45, 44%) but relatively rare among the longer treatment arms.

There was no significant difference between the 36-week and 48-week treatment regimens for the overall cohort. However, among patients with baseline viral load >2 million copies/mL who attained SVR, 65% were treated for 48 weeks and 35% were treated for 36 weeks: all patients with high baseline viral load treated for 24 weeks failed to attain SVR. This suggests that the 48-week treatment regimen may be better suited to patients with high baseline viremia. The efficacy and safety of pegylated interferon 2a has not be adequately evaluated in chronic hepatitis C genotype 4 patients in well conducted clinical trials involving well characterized cohorts and long follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women
2. Age: 25 to 55 years with documented chronic hepatitis
3. Elevated serum alanine aminotransferase at least 2 times the upper limit of normal (40 U/L) on 2 occasions during the preceding 6 months
4. Detectable anti-HCV antibody status assessed by second-generation enzyme-linked immunosorbent assay (Roche Diagnostics, Branchburg, New Jersey); 5. Detectable HCV RNA by polymerase chain reaction (Cobas Amplicor HCV Monitor v2.0 [Roche Diagnostics, Branchburg, New Jersey]; lower limit of quantitation [50 IU/mL])
5. Infection with HCV genotype 4
6. Histologic evidence of chronic hepatitis C in a liver biopsy specimen obtained within the preceding year.

Exclusion Criteria:

1. Hepatitis A, hepatitis B, autoimmune hepatitis, alcoholic liver disease, drug-induced hepatitis.
2. Decompensated liver disease with a history of variceal hemorrhage, ascites, or hepatic encephalopathy.
3. Patients coinfected with schistosomiasis or human immunodeficiency virus
4. leukocyte count lower than 3000 /mm3, neutropenia (<1500 cells/mm3), a hemoglobin level lower than 12 g/dL for women and lower than 13 g/dL for men, thrombocytopenia (<90,000 cells/mm3), creatinine concentration 1.5 times the upper limit of normal
5. Organ transplantation
6. Neoplastic disease
7. Severe cardiac or pulmonary disease
8. Unstable thyroid dysfunction
9. Psychiatric disorder
10. Current pregnancy or breast feeding.
11. Therapy with immunomodulatory agents within the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
SVR, defined as undetectable serum HCV RNA | 24 weeks after discontinuation of treatment

SECONDARY OUTCOMES:
histological response | 24 weeks after completetion of therapy
biochemical response | 24 weeks after therapy completion

CONTACTS AND LOCATIONS:
Overall Officials: Sanaa M Kamal, M.D.; Ph.D, Principal Investigator — Ain Shams University

REFERENCES:
- [Background] Kamal SM, El Tawil AA, Nakano T, He Q, Rasenack J, Hakam SA, Saleh WA, Ismail A, Aziz AA, Madwar MA. Peginterferon alpha-2b and ribavirin therapy in chronic hepatitis C genotype 4: impact of treatment duration and viral kinetics on sustained virological response. Gut. 2005 Jun;54(6):858-66. doi: 10.1136/gut.2004.057182. PMID 15888797
- [Background] El-Zayadi AR, Attia M, Barakat EM, Badran HM, Hamdy H, El-Tawil A, El-Nakeeb A, Selim O, Saied A. Response of hepatitis C genotype-4 naive patients to 24 weeks of Peg-interferon-alpha2b/ribavirin or induction-dose interferon-alpha2b/ribavirin/amantadine: a non-randomized controlled study. Am J Gastroenterol. 2005 Nov;100(11):2447-52. doi: 10.1111/j.1572-0241.2005.00253.x. PMID 16279899
- [Background] Diago M, Hassanein T, Rodes J, Ackrill AM, Sedarati F. Optimized virologic response in hepatitis C virus genotype 4 with peginterferon-alpha2a and ribavirin. Ann Intern Med. 2004 Jan 6;140(1):72-3. doi: 10.7326/0003-4819-140-1-200401060-00035. No abstract available. PMID 14706990
- [Background] Khuroo MS, Khuroo MS, Dahab ST. Meta-analysis: a randomized trial of peginterferon plus ribavirin for the initial treatment of chronic hepatitis C genotype 4. Aliment Pharmacol Ther. 2004 Nov 1;20(9):931-8. doi: 10.1111/j.1365-2036.2004.02208.x. PMID 15521839
- [Derived] Kamal SM, Ahmed A, Mahmoud S, Nabegh L, El Gohary I, Obadan I, Hafez T, Ghoraba D, Aziz AA, Metaoei M. Enhanced efficacy of pegylated interferon alpha-2a over pegylated interferon and ribavirin in chronic hepatitis C genotype 4A randomized trial and quality of life analysis. Liver Int. 2011 Mar;31(3):401-11. doi: 10.1111/j.1478-3231.2010.02435.x. Epub 2011 Jan 11. PMID 21281434